CLINICAL TRIAL: NCT00119171
Title: A Phase I, Open-Label, Dose-Escalation Study of the Safety and Tolerability of Ispinesib in Combination With Capecitabine on an Every 21-Day Schedule in Subjects With Advanced Solid Tumors
Brief Title: Ispinesib In Combination With Capecitabine In Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSP10004
Record Dates: First submitted 2005-07-05; First posted 2005-07-13 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Solid Tumor Cancer
Keywords: Safety; tolerability; dose limiting toxicity; solid tumors; capecitabine
MeSH Terms: interventions — ispinesib; Capecitabine

INTERVENTIONS:
Drug: Ispinesib
Drug: Capecitabine
  Other Names: Ispinesib

SUMMARY:
The purpose of this study is to determine the dose regimen of Ispinesib in combination with capecitabine in patients with solid tumors. Ispinesib is dosed by 1-hour intravenous infusion every 3 weeks and capecitabine is dosed orally, twice a day for 14 days with a 1 week rest period. A patient may continue to receive treatment as long as they are benefiting from the treatment. Blood samples will be taken at specific times to measure the amount of both drugs in your body at specific times after the drug is given. Blood samples will also be taken for lab tests such as complete blood counts and clinical chemistries. Physical exams will be performed before each treatment with Ispinesib. During the treatment phase, the patients will undergo regular assessments for safety and clinical response.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed diagnosis of an advanced solid tumor malignancy that is not responsive to standard therapies or for which there is no standard therapy.
* ECOG (Eastern Cooperative Oncology Group) Performance Status of 0-2.
* Bone marrow function: - ANC greater than 1500/mm3.
* Platelet count greater than or equal to 100,000/mm3.
* Hemoglobin greater than 9 g/dL.
* Renal function: - Calculated creatinine clearance greater than or equal to 50 mL.min.
* Total bilirubin greater than 1.5 mg/dL.
* AST/ALT less than 2.5 X upper limit of normal.

Exclusion criteria:

* Females who are pregnant or nursing.
* Pre-existing hemolytic anemia.
* Pre-existing peripheral neuropathy greater than or equal grade 2.
* Known deficiency in dihydropyrimidine dehydrogenase (DSD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-11

PRIMARY OUTCOMES:
Plasma levels for SB-715992 and Capecitabine | will be checked at Day 1 for Cycle 1.

SECONDARY OUTCOMES:
- Medical history | at screening
- ECOG Performance Status, Physical Exam, vitals, & labs | done at screening, Week 1 (each cycle), & follow-up (f/u)
- Continuous Adverse Event monitoring | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, San Antonio, Texas, United States